CLINICAL TRIAL: NCT02275221
Title: Investigation and Elucidation of Host Immune Responses in Patients With Hepatitic B and C Virus Infection
Brief Title: Immune Response in Patients With Hepatitis B and C Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Other Study IDs: B664
Record Dates: First submitted 2014-10-20; First posted 2014-10-27 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Hepatitis B; Hepatitis C
Keywords: Hepatitis B (HBV); Hepatitis C (HCV)
MeSH Terms: conditions — Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatitis B and C: Hepatitis B and C

SUMMARY:
Using peripheral blood mononuclear cells (PBMC) and serum collection from HBV and HCV infected patients in a number of different immunological assays, the investigators hope to identify any changes in the number and function of these immune cells and to investigate how these changes contribute to viral persistence and disease progression.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) and C (HCV) are the leading causes of liver disease worldwide. Approximately 400 million people worldwide are chronically infected with HBV world wide and it is estimated that 3% of the entire world population is infected with HCV and yet there is still no vaccine available.

Chronic viral hepatitis infection is primarily the result of a complex interaction between the virus and an impaired host immune response. The host immune response has a unique role in HBV and HCV infection because it contributes not only to viral control clinical recovery and protective immunity but also to the development of chronic hepatitis and liver cirrhosis. There is currently no cure for most patients who already have chronic HBV and HCV infection and a proportion of patients fail to respond to current antiviral regimens. Since these patient remain at risk for disease progression it is crucial to investigate host immune responses and to determine the precise role of these responses in disease outcome.

Using peripheral blood mononuclear cells (PBMC) and serum collection from HBV and HCV infected patients in a number of different immunological assays, we hope to identify any changes in the number and function of these immune cells and to investigate how these changes contribute to viral persistence and disease progression. This information can be utilised to develop more effective treatment regimens in order to reduce the current global burden of these diseases.

ELIGIBILITY:
Inclusion Criteria:

Chronic Hepatitis B patients At all stages of infection Treatment naive and previously treated Longitudinal samples from patients treated with antiviral agents and interferon

Chronic Hepatitis C patients All genotypes - treatment naive and previously treated Longitudinal samples from patients treated with interferon and STATIC therapy

Exclusion Criteria:

Coinfection with HIV Coinfection with hepatitis delta Excessive alcohol use Autoimmune liver disease Metabolic liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis B and C
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To investigate whether changes in immune cell response for in-patients with Hepatitis B or C can be used to develop better treatment regimes | on average 4 weeks
  The principle aim of this study is to investigate exactly how patients; immune cells interact with hepatitis B and C virus after becoming infected. By understanding how the immune cells interact with the virus it will be possible to use this information to develop better treatment regimens for these patients

SECONDARY OUTCOMES:
Changes in immune cell reaction as determined by cytokine expression for patients with Hepatitis B during their inpatient stay | on average 4 weeks
  During their in-patient stay patients with Hepatitis B will have their cytokine expression recorded to determine whether this has an effect on their immune cell response
Changes in immune cell reaction as determined by cytokine expression for patients with Hepatitis C during their inpatient stay | on average 4 weeks
  During their in-patient stay patients with Hepatitis C will have their cytokine expression recorded to determine whether this has an effect on their immune cell response
Changes in immune cell reaction as determined by t-cell populations for patients with Hepatitis B during their inpatient stay | on average 4 weeks
  During their in-patient stay patients with Hepatitis B will have their t-cell populations recorded to determine whether this has an effect on their immune cell response
Changes in immune cell reaction as determined by t-cell populations for patients with Hepatitis C during their inpatient stay | on average 4 weels
  During their in-patient stay patients with Hepatitis C will have their t-cell populations recorded to determine whether this has an effect on their immune cell response

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Wright, MBBS MRCP, Principal Investigator — Basildon and Thurrock University Hospitals NHS FT
Locations (1):
- Basildon Hospital, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No